CLINICAL TRIAL: NCT01535274
Title: The Influence of Basic Ventilation Strategies and Anesthetic Techniques on Cerebral Oxygenation in the Beach Chair Position
Brief Title: Ventilation Strategies, Anesthetic Techniques and Cerebral Oxygenation in the Beach Chair Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Paul Picton, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00049747
Record Dates: First submitted 2012-02-09; First posted 2012-02-17 (Estimated); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: Cerebral oxygenation; Beach chair position; General anesthetic technique; Inspired oxygen fraction; End tidal carbon dioxide
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desflurane (Experimental): Patients will receive general anesthesia with desflurane. Both arms have rSO2 measured and undergo identical changes in ventilation strategy.
  Interventions: Other: Inspired oxygen fraction / end tidal carbon dioxide
- Propofol (Experimental): Patients will receive total intravenous general anesthesia (TIVA) with propofol. Both have rSO2 measured and undergo identical changes in ventilation strategy.
  Interventions: Other: Inspired oxygen fraction / end tidal carbon dioxide

INTERVENTIONS:
Other: Inspired oxygen fraction / end tidal carbon dioxide — Following induction of anesthesia, FIO2 and minute ventilation will be sequentially adjusted to achieve:
  1. FIO2 30% (70% nitrogen), PETCO2 30mmHg - supine position.
  2. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
  3. FIO2 100%, PETCO2 30mmHg - beach chair position.
  4. FIO2 100%, PETCO2 45mmHg - beach chair position.
  5. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.

SUMMARY:
The seated or "beach chair" position during surgery and general anesthesia decreases brain oxygen levels and can result in stroke. As such, poor neurological outcome following beach chair positioning is a growing concern. In the proposed study the investigators test the hypothesis that changes in ventilation strategy and anesthetic technique can affect cerebral oxygenation in anesthetized patients in the beach chair position.

DETAILED DESCRIPTION:
This is a prospective cohort study with randomized nested design. Patients presenting for shoulder surgery will be randomized to receive desflurane or total intravenous anesthesia with propofol. Regional cerebral oxygenation will be measured using the INVOS 5100C monitor (Covidien, Boulder, CO). Depth of anesthesia will be maintained within a Bispectral Index range of 40-60. Following positioning, inspired oxygen fraction and minute ventilation will be sequentially adjusted. At each set point, regional cerebral oxygenation will be recorded and venous blood gas analysis performed. Statistical analysis will be repeated measures analysis of variance in which ventilation strategy is the within-subjects factor and anesthetic technique is the between-subjects factor; post hoc Tukey's correction will be used for multiple comparisons. If simple maneuvers of ventilation and anesthetic technique can prevent low brain oxygen levels, patient outcome may be improved.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective arthroscopic shoulder surgery in the beach chair position under general anesthesia with supplemental interscalene block

Exclusion Criteria:

* refusal to give consent
* ineligible for interscalene block
* history of cardiovascular disease
* history of cerebrovascular disease
* hypertension
* respiratory failure
* non-English speaker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Picton, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Picton P, Dering A, Miller B, Shanks A, Mashour GA. The influence of basic ventilation strategies and anesthetic techniques on cerebral oxygenation in the beach chair position: study protocol. BMC Anesthesiol. 2012 Sep 20;12:23. doi: 10.1186/1471-2253-12-23. PMID 22994896

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten potential participants were excluded for not meeting inclusion criteria, declination to participate, and other reasons.
Groups:
- Propofol: Patients received total intravenous general anesthesia (TIVA) with propofol. Both have rSO2 measured and undergo identical changes in ventilation strategy.
  Inspired oxygen fraction / end tidal carbon dioxide: Following induction of anesthesia, FIO2 and minute ventilation was sequentially adjusted to achieve:
  1. FIO2 30% (70% nitrogen), PETCO2 30mmHg - supine position.
  2. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
  3. FIO2 100%, PETCO2 30mmHg - beach chair position.
  4. FIO2 100%, PETCO2 45mmHg - beach chair position.
  5. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
- Desflurane: Patients received general anesthesia with desflurane. Both arms have rSO2 measured and undergo identical changes in ventilation strategy.
  Inspired oxygen fraction / end tidal carbon dioxide: Following induction of anesthesia, FIO2 and minute ventilation was sequentially adjusted to achieve:
  1. FIO2 30% (70% nitrogen), PETCO2 30mmHg - supine position.
  2. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
  3. FIO2 100%, PETCO2 30mmHg - beach chair position.
  4. FIO2 100%, PETCO2 45mmHg - beach chair position.
  5. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
Period: Overall Study
Arm/Group | Propofol | Desflurane
Started | 28 | 29 (29 participants were initially randomized to receive desflurane treatment. One participant initially randomized to the desflurane arm was misallocated to the propofol arm and received propofol treatment, as shown in the "reason not completed" section below.)
Received Propofol | 28 | 1 (Of the 29 participants initially randomized to receive desflurane treatment, one was misallocated to the propofol arm and received propofol treatment, as shown in the "reason not completed" section below. That participant is included in the baseline characteristics, outcome measures, and adverse events with the propofol arm.)
Received Desflurane | 0 | 28
Completed | 28 | 27
Not Completed | 0 | 2
Not completed — Determined to be ineligible | 0 | 1
Not completed — Misallocated to propofol intervention | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the 29 participants were initially randomized to receive Desflurane treatment, one misallocated to the Propofol arm and received Propofol treatment, and is included in the propofol arm for baseline measure for that reason.
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Desflurane | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (10.0) | 49.3 (13.3) | 50.34 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 18 | 17 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Regional Cerebral Oxygenation (rSO2) Before and 5 Minutes After Each Change in Ventilation Strategy
Description: rSO2 will be recorded as a "snap shot." A mean value from right and left sides will be calculated for each patient at each study point.
  Set Point 1: FIO2 30% (70% nitrogen), PETCO2 30mmHg - supine position. Set Point 2: FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position. Set Point 3: FIO2 100%, PETCO2 30mmHg - beach chair position. Set Point 4: FIO2 100%, PETCO2 45mmHg - beach chair position. Set Point 5: FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
  With each set point, the value shown is the absolute change from baseline.
Time Frame: duration of surgery, generally no more than 90 minutes total
Population: Of the 29 participants initially randomized to receive desflurane treatment, one participant initially randomized to the desflurane arm was misallocated to the propofol arm and received propofol treatment, so is included in the propofol arm here.
Measure: Mean (Standard Deviation); unit: Percent oxygen saturation
Arm/Group | Propofol | Desflurane
Number analyzed (Participants) | 29 | 27
Percent oxygen saturation
  Set Point 1: FIO2 30%; PETCO2 30mmHg (Supine) | -4.27 (8.43) | -0.70 (10.08)
  Set Point 2: FIO2 30%; PETCO2 30mmHg (Beach Chair) | -15.48 (11.35) | -10.90 (7.03)
  Set Point 3: FIO2 100%; PETCO2 30mmHg (Beach Chair) | -8.31 (11.21) | -3.14 (7.21)
  Set Point 4: FIO2 100%; PETCO2 45mmHg (Beach Chair) | 5.46 (9.79) | 9.20 (7.01)
  Set Point 5: FIO2 30%; PETCO2 30mmHg (Beach Chair) | -9.00 (11.02) | -3.59 (7.67)

2. Primary Outcome: Regional Cerebral Oxygenation (rSO2) Values
Description: Regional cerebral oxygenation (rSO2) values at the set ventilatory points of the study for each anesthetic choice.
  Set Point 1: FIO2 30% (70% nitrogen), PETCO2 30mmHg - supine position. Set Point 2: FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position. Set Point 3: FIO2 100%, PETCO2 30mmHg - beach chair position. Set Point 4: FIO2 100%, PETCO2 45mmHg - beach chair position. Set Point 5: FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
Time Frame: duration of surgery, generally no more than 90 minutes total
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage cerebral oxygen saturation
Groups:
- Propofol: Patients will receive total intravenous general anesthesia (TIVA) with propofol. Both have rSO2 measured and undergo identical changes in ventilation strategy.
  Inspired oxygen fraction / end tidal carbon dioxide: Following induction of anesthesia, FIO2 and minute ventilation will be sequentially adjusted to achieve:
  1. FIO2 30% (70% nitrogen), PETCO2 30mmHg - supine position.
  2. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
  3. FIO2 100%, PETCO2 30mmHg - beach chair position.
  4. FIO2 100%, PETCO2 45mmHg - beach chair position.
  5. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
- Desflurane: Patients will receive general anesthesia with desflurane. Both arms have rSO2 measured and undergo identical changes in ventilation strategy.
  Inspired oxygen fraction / end tidal carbon dioxide: Following induction of anesthesia, FIO2 and minute ventilation will be sequentially adjusted to achieve:
  1. FIO2 30% (70% nitrogen), PETCO2 30mmHg - supine position.
  2. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
  3. FIO2 100%, PETCO2 30mmHg - beach chair position.
  4. FIO2 100%, PETCO2 45mmHg - beach chair position.
  5. FIO2 30% (70% nitrogen), PETCO2 30mmHg - beach chair position.
Arm/Group | Propofol | Desflurane
Number analyzed (Participants) | 29 | 27
Percentage cerebral oxygen saturation
  Set Point 1: Fio2 0.3 Petco2 30 mmHg | 67 (13) | 69 (11)
  Set Point 2: Fio2 0.3 Petco2 30 mmHg | 59 (13) | 62 (10)
  Set Point 3: Fio2 1.0 Petco2 30 mmHg | 64 (14) | 67 (11)
  Set Point 4: Fio2 1.0 Petco2 45 mmHg | 74 (12) | 76 (11)
  Set Point 5: Fio2 0.3 Petco2 30 mmHg | 64 (14) | 67 (12)
Statistical Analysis 1: Comparison: Propofol vs Desflurane; P-values represent comparison of successive set points within anesthetic type (i.e.: Set Point 1 compared to Set Point 2, Set Point 2 compared to Set Point 3, etc.). This P-value was determined for each of set points 1, 2, 3, 4, and 5; Test type: Superiority; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: During the time of surgery - not more than 90 minutes
Description: Study team used a non-systematic approach for collecting adverse event information, reliant on patient self-reporting and study team observation during treatment.
Arm/Group | Propofol | Desflurane
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes